CLINICAL TRIAL: NCT03695861
Title: Contribution of 18F-FDG PET-CT in the Diagnosis and the Detection of Peripheral Emboli of Infectious Endocarditis on Native Valves
Acronym: NATIVTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2017/33
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Endocarditis
Keywords: Endocarditis Infectious; Native valve; ESC 2015 modified diagnostic criteria; 18F-FDG PET-CT; Detection of peripheral emboli
MeSH Terms: conditions — Endocarditis; Endocarditis, Subacute Bacterial

STUDY DESIGN:
Intervention Model Description: Diagnostic study, prospective, "delayed-type cross-sectional study" (the result of the reference test is defined at 3 months of follow-up), monocentric, blinded, including consecutive patients.
Masking Description: The interpretation of the PET-CT will be performed by a nuclear medicine expert who is expert in cardiac imaging and infectious pathology, blinded to other imaging tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole-body 18F-FDG PET-CT scan (Experimental)
  Interventions: Diagnostic Test: Whole-body 18F-FDG PET-CT scan

INTERVENTIONS:
Diagnostic Test: Whole-body 18F-FDG PET-CT scan — A 18F-FDG PET-CT will be performed within 5 days of the beginning of the patients care with infectious endocarditis at the University Hospital center of Bordeaux.

SUMMARY:
The diagnosis of infectious endocarditis is not always easy and is based on several clinical and imaging arguments. Positron Emission Tomography - Computed Tomography (PET-CT) has been validated for endocarditis on prosthetic valves but few studies concern the native valves. The purpose of the study is to estimate the diagnostic sensitivity of [18F]-fluoro-2-deoxyglucose (18F-FDG) PET-CT in patients with endocarditis on native valves according to the European Society of Cardiology 2015 (ESC 2015) modified diagnostic criteria of infective endocarditis classified as definite at three months of follow-up (baseline test).

DETAILED DESCRIPTION:
Infectious endocarditis remains a serious pathology with an intra-hospital mortality of between 15 and 30%. The prognosis of patients depends on the speed of diagnosis and the beginning of the appropriate treatment.

Currently, the diagnosis of endocarditis is based on the ESC 2015 modified criteria. Echocardiography techniques play a key role, but can be negative in 20% of endocarditis. 18F-FDG PET-CT showed promising results in the management of prosthetic valve endocarditis and / or stimulation material.

However, few studies have been carried out on the contribution of PET-CT in the diagnosis of endocarditis on native valves, with discordant results. But this is the majority of endocarditis (70% of cases).

A 18F-FDG PET-CT will be performed in all patients included in the study in addition to standard care for endocarditis, within 5 days of the beginning of their management in the university hospital center of Bordeaux after verification of inclusion and exclusion criteria and signature of consent.

The included patients will be reviewed at Month 3 during a consultation with the completion of a clinical examination, an electrocardiogram, a biological assessment and a transthoracic ultrasound.

Adverse events and serious adverse events will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ≥ 18 years treated at the university hospital center of Bordeaux for suspicion of infectious endocarditis on a native valve with a "definite" or "possible" diagnosis according to the ESC 2015 modified diagnostic criteria, agreeing to participate,
* Affiliated person or beneficiary of a social security scheme,
* Free, informed and written consent (no later than the day of inclusion and before any exam required by the research).

Exclusion Criteria:

* Patient with a vital failure (haemodynamic, respiratory or neurological instability), requiring treatment in the intensive care unit and / or urgent surgery incompatible with performing PET-CT,
* Pregnant or nursing woman,
* Patient who has already been treated for infective endocarditis within six months of enrollment,
* Patient who had cardiac surgery in the two months preceding inclusion,
* Patient who has previously been hypersensitive to fluorodeoxyglucose and / or excipients of the radiotracer,
* Patient unable to sign consent,
* Patient under legal protection,
* Women of childbearing age who do not benefit from effective contraception (HAS criteria),
* Patient in a period of relative exclusion from another research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the 18F-FDG PET-CT in the diagnosis of infectious endocarditis | 3 month
  The reference test in this study will be a "definite diagnosis" of infectious endocarditis according to the ESC 2015 modified criteria at three months of follow-up, evaluated by a multidisciplinary committee in infectious endocarditis. This evaluation will be done blind to the results of the PET-CT of the study. The index test 18F-FDG PET-CT will have been performed at the initial phase of patient management.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile ALEXANDRINO, MD, Principal Investigator — University Hospital, Bordeaux; Paul PEREZ, MD,PhD, Study Chair — University Hospital, Bordeaux
Locations (1):
- University hospital, Bordeaux, Pessac, France